CLINICAL TRIAL: NCT04990726
Title: Immune Related Toxicity and Symptom Burden in Chronic Cancer Survivors With Melanoma Receiving Adjuvant Immunotherapy With Immune Checkpoint Inhibitors
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0390; NCI-2020-13274 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0390 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-02-11; First posted 2021-08-04 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Clinical Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage III Cutaneous Melanoma AJCC v8; Pathologic Stage IIIA Cutaneous Melanoma AJCC v8; Pathologic Stage IIIB Cutaneous Melanoma AJCC v8; Pathologic Stage IIIC Cutaneous Melanoma AJCC v8; Pathologic Stage IIID Cutaneous Melanoma AJCC v8; Melanoma, Stage II; Melanoma Stage IV
MeSH Terms: conditions — Melanoma | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Observational (assessment, blood collection, questionnaire): Patients undergo medical assessments and blood sample collection and complete questionnaires at baseline, 1, 3, 6, 12, 18, and 24 months.
  Interventions: Behavioral: Assessment; Procedure: Biospecimen Collection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Treatment (assessment, blood collection, questionnaire): Patients undergo medical assessments and blood sample collection and complete questionnaires at baseline (prior to C1 infusion), 2, 4, 7 infusion, at end of treatment, and 18 and 24 months after completion of treatment.
  Interventions: Behavioral: Assessment; Procedure: Biospecimen Collection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Assessment — Undergo medical assessments
  Other Names: Assess
Procedure: Biospecimen Collection — Undergo collection of blood samples
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study evaluates the immune related toxicity and symptom burden in chronic cancer survivors with melanoma who are receiving adjuvant immunotherapy with immune checkpoint inhibitors. Information collected in this study may help doctors to learn more about the side effects caused by immunotherapy, and to learn if there are any relationships between these side effects and immune and genetic biomarkers found in the blood that may be related to patient's reaction to immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the detailed clinical characterization including timing, severity, and phenotype of immune related adverse events (irAEs) in chronic survivors with melanoma from initiation of adjuvant checkpoint inhibitors (CPI) therapy through 24 months of follow-up.

II. Longitudinally assess patients-reported outcomes (PROs) that measure symptom burden (such as fatigue, depression, sleep disturbance) and quality of life (QOL) in those patients, compared to patients with similar disease stage who opt for active surveillance.

SECONDARY OBJECTIVES:

I. Longitudinally evaluate the correlation of changes in immune analysis (immune cells and cytokines) in peripheral blood samples with timing, severity, and phenotype of irAEs, symptom burden, and QOL in those patients, compared to patients with similar disease stage who opt for active surveillance.

II. Determine whether specific immune-related genetic polymorphisms are associated with the development of irAEs and symptom burden in melanoma patients receiving adjuvant CPI therapy.

OUTLINE:

Patients undergo medical assessments and blood sample collection, and complete questionnaires at baseline, 1 (optional), 3, 6, 12, 18, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years of age
* Surgically resected stage II, III, or IV melanoma with no evidence of disease according to the American Joint Committee on Cancer (AJCC) classification criteria
* Eligible for adjuvant CPI treatment per treating physician discretion
* Plan to continue care at MD Anderson Cancer Center (MDACC)
* Ability to communicate and read in English language

Exclusion Criteria:

* Previous systemic therapy for melanoma
* Previous history of other cancers treated with immunotherapy

  * Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
  * Previous cancer that has been resected two or more years ago are not excluded.
* Previous history of inflammatory or autoimmune diseases. This include but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or psoriasis. Patients with autoimmune thyroid disease, vitiligo, and type I diabetes mellitus are not excluded.
* Other concurrent malignancies that require active therapy
* Participants < 18 years of age and pregnant women are not eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with resected melanoma who are eligible for adjuvant CPI treatment
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Detailed clinical characterization | 24 months
  Will determine the detailed clinical characterization including timing, severity, and phenotype of immune related adverse events (irAEs) in chronic survivors with melanoma from initiation of adjuvant checkpoint inhibitor (CPI) therapy through 24 months of follow-up. The primary end point will be at 12 months, but patients will be followed for up to 24 months. Will estimate the incidence rates of any de novo grade 2 or higher irAEs at 12 months post treatment initiation along with 95% confidence interval within the case group. Will also summary irAEs by their onset time in relation to treatment initiation (acute irAE vs late irAE) and by CPI type. Descriptive statistics will be used to summarize results.
Patients-reported outcomes (PROs) | 24 months
  Will compare PROs at 12 months between the case (with and without irAEs) and control groups. To compare differences between cases and controls, will use logistic regression to adjust for age, gender, ethnicity, tumor stage and type of CPI therapy. The primary outcome measures include quality of life, depression, and fatigue. Will compare each of the three primary outcomes at a significant level of 0.017 (0.05/3) using Bonferroni multiple comparison adjustment. Will use linear mixed effect models to fit the longitudinal PRO assessments to study the change of PROs over time taking the intra-patient correlation into account and to determine the effect of each of the covariates (relevant patient's demographic, irAEs, clinical and treatment characteristics) on the outcomes.

SECONDARY OUTCOMES:
Changes in immune analysis | 24 months
  Will longitudinally evaluate the correlation of changes in immune analysis in peripheral blood samples with timing, severity, and phenotype of irAEs, symptom burden, and quality of life in those patients, compared to patients with similar disease stage who opt for active surveillance.
Immune-related genetic polymorphisms | 24 months
  Will determine whether specific immune-related genetic polymorphisms are associated with the development of irAEs and symptom burden in melanoma patients receiving adjuvant CPI therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Noha Hassan, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org